CLINICAL TRIAL: NCT01296204
Title: Phase I of Radioimmunotherapy (RIT) in MULTIPLE MYELOMA Using the Antibody B-B4 Radiolabelled With IODE 131
Brief Title: Radioimmunotherapy (RIT) in MULTIPLE MYELOMA Using the Antibody B-B4 Radiolabelled With IODE 131
Acronym: BB4
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Centre René Gauducheau (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 04/1B
Record Dates: First submitted 2011-02-11; First posted 2011-02-15 (Estimated); Last update posted 2011-03-22 (Estimated); Status verified 2011-02

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- BB4 antibody-Iodine 131 (Experimental)
  Interventions: Drug: BB4 antibody-Iodine 131

INTERVENTIONS:
Drug: BB4 antibody-Iodine 131 — Injection of an antibody after labelling with Iodine 131

SUMMARY:
The first step of this protocol called step pre-treatment study the biodistribution and pharmacokinetics of a tracer dose of radiolabeled antibody. The second step called step therapy study the toxicity and antitumor effects of antibody B-B4 coupled with increasing doses of iodine 131. At least 17 patients will be included for an estimated duration of 2 years to determine the maximum tolerated dose and dose limiting toxicity. The immediate side effects, medium and long terms will be analyzed. After determining the toxic dose limit, patients will be treated at the maximum tolerated dose, for a total of 15 patients at this level, which will measure the objective tumor response to treatment. These patients will be followed for 1 year after injection therapy.

ÉcouterLire phonétiquement

ELIGIBILITY:
Inclusion Criteria:

* Patients with a confirmed diagnosis of multiple myeloma (> 10% plasma cells on a previous myelogram)
* Secretion of a monoclonal immunoglobulin
* No myelodysplasia evaluated by myelogram
* Disease refractory or relapsed after at least 3 lines of therapy
* Patients with a dated and signed the consent form
* Collection of autologous peripheral blood stem cells containing at least 2. 106 CD 34 + cells / kg
* Age> 18 years
* Performance status <2 (see Annex I), life expectancy of more than 3 months
* No chemotherapy or radiotherapy within 4 weeks before inclusion
* No major surgery within 4 weeks preceding the assessment of inclusion
* No bisphosphonates within 2 weeks prior radioimmunotherapy, except for treatment started more than three months ago.
* Normality of the biological assessment:
* Creatinine less than or equal to 1.5 times the normal laboratory
* Liver: less than or equal to 1.5 times the normal laboratory (free and conjugated bilirubin, SGOT, SGPT, gamma GT PAL)
* Hemoglobin ≥ 8 g/mm3
* ≥ 3 WBC 000/mm3
* Neutrophils ≥ 1 500/mm3
* Platelets ≥ 100 000/mm3

Exclusion Criteria:

Patients with other cancers except uterine carcinoma in situ or basal cell skin carcinoma

* Patients with other (s) condition (s) Severe (s) to prevent tolerance to study and conduct the study to completion
* Patient is pregnant or unwilling to take a contraceptive treatment for three months after treatment
* Collection of peripheral blood stem cells containing less than 2106 CD 34 + cells / kg
* Patients enrolled in another experimental treatment protocol
* Patients who already received treatment with radioimmunotherapy
* Myelodysplasia assessed by myelogram
* Patient with thyroid
* Patient unable to sign informed consent ÉcouterLire phonétiquement

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33

PRIMARY OUTCOMES:
The dose limiting toxicities (DLT) will be analysed in order to determine the maximal tolerated dose (MTD) in a dose escalation study design.

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Centre René Gauducheau, Nantes
  - Moreau, Nantes